CLINICAL TRIAL: NCT02228681
Title: A Randomized Phase II Trial of Everolimus and Letrozole or Hormonal Therapy (Tamoxifen/Medroxyprogesterone Acetate) in Women With Advanced, Recurrent, or Persistent Endometria Carcinoma
Brief Title: Everolimus and Letrozole or Hormonal Therapy to Treat Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3007; CRAD001CUS236T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2014-08-14; First posted 2014-08-29 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Advanced, Persistent, or Recurrent Endometrial Cancer
MeSH Terms: interventions — Everolimus; Tamoxifen; Letrozole; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus and Letrozole (Experimental): Everolimus 10 mg daily and Letrozole 2.5 mg PO daily
  Interventions: Drug: Everolimus; Drug: Letrozole
- Hormonal Therapy (Active Comparator): Tamoxifen 20 mg PO BID; on alternating weeks (even numbered) weeks, Medroxyprogesterone Acetate 200 mg PO daily with Tamoxifen 20 mg PO BID
  Interventions: Drug: Tamoxifen; Drug: Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Everolimus — 10mg daily by mouth
  Other Names: RAD001
  Arms: Everolimus and Letrozole
Drug: Tamoxifen — 20 mg daily by mouth on alternating weeks (even numbered) weeks
  Other Names: Nolvadex®
  Arms: Hormonal Therapy
Drug: Letrozole — 2.5mg once a day by mouth
  Other Names: Femara®
  Arms: Everolimus and Letrozole
Drug: Medroxyprogesterone Acetate — 200 mg daily by mouth
  Arms: Hormonal Therapy

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of the combination of the drugs Everolimus and Letrozole compared to Tamoxifen and Medroxyprogesterone acetate in treating endometrial cancer and to determine the types and severity of side effects caused by treatment with these drug combinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced (FIGO Stage III or IV), persistent, or recurrent endometrial carcinoma, which is not likely to be curable by surgery or radiotherapy. Histologic documentation of the recurrence is not required.
* All patients must have measurable disease. Measurable disease is defined by RECIST version 1.1). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be greater than or equal to 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or greater than or equal to 20 mm when measured by chest x-ray. Lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI (See section 8).
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1 (Section 8.1). Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* Prior chemoradiotherapy for a pelvic recurrence is permitted. Prior chemotherapy in the adjuvant setting for Stage I, II or III disease is permitted.

Note: No prior chemotherapy in the setting of Stage IV disease is permitted unless the patient was without evidence of disease at the completion of chemotherapy and had at least six months of progression-free survival since the completion of chemotherapy.

Regardless of circumstances, no more than one prior chemotherapy regimen (including chemo-radiotherapy) is permitted.

* Patient must be able to take p.o. medications.
* Performance status must be 0-1.
* Patients must have adequate organ and marrow function as defined below:

NOTE: Institutional/laboratory upper limit of normal = ULN Institutional/laboratory lower limit of normal = LLN

* Bone marrow function:

  * Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
  * Platelets greater than or equal to 100,000 cells/mcl
  * Hemoglobin greater than or equal to 9 g/dL
* Coagulation

  • INR less than or equal to 1.5 x ULN (or in range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin).
* Renal function:

  • Creatinine less than or equal to 1.5 x ULN
* Hepatic function:

  * Bilirubin less than or equal to 1.5 x ULN
  * ALT and AST less than or equal to 3 x ULN
  * Alkaline phosphatase less than or equal to 2.5 x ULN
  * Albumin greater than or equal to 2.8 g/dL
* Lipid panel:

  * Fasting serum cholesterol less than or equal to 300 mg/dL
  * Fasting triglycerides less than or equal to 300 mg/
* At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: hysterectomy, resection of a lung nodule; minor: central venous access catheter placement).
* At least 4 weeks must have elapsed since the patient received any radiation therapy.
* Patients who have met the pre-entry requirements specified in Section 7.0
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* All patients must be at least 18 years of age
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing a highly effective form of contraception.

During the study treatment and for 8 weeks after stopping the treatment. Highly effective contraception methods include combination of any two of the following:

* Use of oral, injected or implanted hormonal methods of contraception or;
* Placement of an intrauterine device (IUD) or intrauterine system (IUS);
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
* Total abstinence or;
* Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.

Exclusion Criteria:

* Patients who have previously received everolimus, any another mTOR inhibitor or any agent targeting the PI3K/AKT/mTOR pathway.
* Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Patients who have previously received hormonal therapy for endometrial cancer.
* Patients with concomitant invasive malignancy or a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the past five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol.
* Patients receiving chronic treatment with systemic steroids or another immunosuppressive agent.
* Patients with active or uncontrolled systemic infection.
* Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and anti-diabetic treatment must be monitored closely throughout the trial and adjusted as necessary.
* Known severely impaired lung function, including:

  • CTCAE grade 2 (or greater) hypoxia (decreased oxygen saturation with exercise [e.g., pulse oximeter <88%]; intermittent supplemental oxygen)
* Patients with a known history of cardiac disease. This includes:
* Uncontrolled hypertension, defined as systolic greater than 150 mm Hg or diastolic greater than 90 mm Hg despite antihypertensive medications.
* Myocardial infarction or unstable angina within 6 months prior to registration.
* New York Heart Association (NYHA) Class II or greater congestive heart failure.
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or serious cardiac arrhythmia requiring medication. This does not include asymptomatic atrial fibrillation with controlled ventricular rate.
* Cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) within 6 months prior to the first date of study therapy.
* Patients who are pregnant or breast-feeding.
* Patients with known central nervous system metastases.
* Patients with known human immunodeficiency virus (HIV) infection.
* Patients with an impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease; uncontrolled nausea, vomiting and/or diarrhea; malabsorption syndrome; clinical signs and symptoms of gastrointestinal obstruction; and/or patients who require parenteral hydration and/or nutrition).
* Patients who plan to receive live attenuated vaccines within 1 week of start of everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder or coagulopathy.
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 30 days prior to dosing.
* Patients must be able to follow concomitant medication restrictions:

  * Avoid the use of strong CYP3A/PgP inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, indinavir, nelfinavir, voriconazole).
  * Use caution when co-administered with moderate CYP3A4/PgP inhibitors (e.g., amprenavir, fosamprenavir, aprepitant, erythromycin, fluconazole, verapamil, diltiazem).
  * Grapefruit, grapefruit juice, and other foods known to inhibit cytochrome P450 and PgP activity may increase everolimus exposures and should be avoided during treatment.
  * Avoid the use of concomitant strong CYP3A4/PgP inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, and phenobarbital).
  * St. John's Wort may decrease everolimus exposure unpredictably and should be avoided.
* Patients with active hepatitis B or C. Screening for hepatitis B

Prior to randomization/start of everolimus, the following three categories of patients should be tested for hepatitis B viral load and serologic markers, that is, HBsAg, HBcAb, HBsAb and quantitative hepatitis B DNA PCR (HBV-DNA):

• All patients who currently live in (or have lived in) Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal and Greece.

[http://wwwnc.cdc.gov/travel/yellowbook/2012/chapter-3-infectious-diseases-related-to-travel/hepatitis-b.htm]

* Patients with any of the following risk factors:
* known or suspected past hepatitis B infection,
* blood transfusion(s) prior to 1990,
* current or prior IV drug users,
* current or prior dialysis,
* household contact with hepatitis B infected patient(s),
* current or prior high-risk sexual activity,
* body piercing or tattoos,
* mother known to have hepatitis B
* history suggestive of hepatitis B infection, e.g., dark urine, jaundice, right upper quadrant pain.
* Additional patients at the discretion of the investigator The management guidelines, in Section 6, are provided according to the results of the baseline assessment of viral load and serological markers for hepatitis B.

Screening for hepatitis C

Patients with any of the following risk factors for hepatitis C should be tested using quantitative RNA-PCR:

* known or suspected past hepatitis C infection (including patients with past interferon 'curative' treatment),
* blood transfusions prior to 1990,
* current or prior IV drug users,
* current or prior dialysis,
* household contact of hepatitis C infected patient(s),
* current or prior high-risk sexual activity,
* body piercing or tattoos. At the discretion of the investigator, additional patients may also be tested for hepatitis C.

The management guidelines, in Section 6 are provided according to the results of the baseline assessment of hepatitis C viral load.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Slomovitz, MD, Study Chair — Gynecologic Oncology Group
Locations (26):
- United States (26):
  - University of Colorado - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Maine Medical Center, Scarborough, Maine
  - Johns Hopkins, Baltimore, Maryland
  - University of Massachusetts Memorial Center, Worcester, Massachusetts
  - Sanford Clinic North - Bemidji, Bemidji, Minnesota
  - St. Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - New Mexico Cancer Alliance, Albuquerque, New Mexico
  - Memorial Medical Center-Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Sanford Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 02/19/2015 and closed to accrual on 04/18/2016. All patients underwent disease evaluation and were found to have measurable histologically confirmed advanced stage, persistent or recurrent endometrial carcinoma. After obtaining informed consent and verification of eligibility, patients were enrolled and treated.
Groups:
- Everolimus and Letrozole: Everolimus 10 mg daily plus letrozole 2.5 mg PO daily in a 28 day cycle.
- Tamoxifen and Medroxyprogesterone Acetate: Tamoxifen 20 mg PO bid days 1-28 plus medroxyprogesterone acetate 200 mg PO days 8-14 and 22-28 repeating in a 28 day cycle.
Period: Overall Study
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.1) | 66.8 (7.3) | 65 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 32 | 31 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Response
Description: A confirmed complete or partial response as defined by RECIST 1.1 was considered a response. "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From date of randomization until the date of first documented progression or date of death , up to 3 years.
Population: Eligible and treated participants. One participant in arm II was not treated. Participant flow contains all eligible participants.
Measure: Number; unit: Number of participants
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate
Number analyzed (Participants) | 37 | 36
Number of participants | 9 | 8

2. Secondary Outcome: Median Progression-free Survival
Description: Progression-free Survival is defined as the duration alive from study entry until progression is documented, or death; whichever comes sooner. Progressive disease is defined as at least a 5 mm absolute increase and a 20% relative increase in the sum of measurable target lesions' longest dimensions relative to the smallest sum at baseline or on study or the appearance of new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Tumor measurements were done at 8 and 16 weeks after initiating treatment and then every 12 weeks and compared with baseline measurements prior to treatment. Measurements are continued until disease progression is documented or death.
Population: Eligible Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate
Number analyzed (Participants) | 37 | 37
months | 6.4 [3.8 to 17.7] | 3.7 [2.5 to 8.9]

3. Secondary Outcome: Frequency and Severity of CTCAE (Common Toxicity Criteria for Adverse Events) Version 4
Description: Maximum grade of physician assessed adverse events graded and categorized using Common Toxicity Criteria for Adverse Events (CTCAE) version 4
Time Frame: Assessed throughout the treatment period and for 30 days after discontinuation of treatment. Treatment continues until progression of disease.
Population: Eligible and Treated Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate
Number analyzed (Participants) | 37 | 36
Participants
  Grade 1 | 2 | 2
  Grade 2 | 6 | 14
  Grade 3 | 27 | 17
  Grade 4 | 2 | 2
  Grade 5 | 0 | 1

4. Secondary Outcome: Median Survival
Description: Survival is defined as the duration alive from study entry until death.
Time Frame: Following treatment discontinuation, patients are followed quarterly for 2 years, semi-annually for 3 more years, annually thereafter.
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate
Number analyzed (Participants) | 37 | 37
Months | NA [14.2 to NA] — No upper limit or median estimate can be provided as the median survival time has not been reached. | 16.6 [7.6 to NA] — No upper limit or median estimate can be provided as the median survival time has not been reached.

5. Other Pre Specified Outcome: Hormone Receptor Immunohistochemistry
Description: To determine if relevant biomarkers correlate with response to treatment in each of the two arms. Unstained sections of tumor tissue will be used for hormone receptor (estrogen receptor-alpha, estrogen receptor-beta, progesterone receptor-A, progesterone receptor B and the G protein-coupled estrogen receptor, GPR-30) immunohistochemistry.
Time Frame: At study entry
Reporting Status: Not Posted

6. Other Pre Specified Outcome: mTOR Pathway Immunohistochemistry
Description: To determine if relevant biomarkers correlate with response to treatment in each of the two arms. Unstained sections of tumor tissue will be used for mTOR pathway (including phosphorylated S6 ribosomal protein, PTEN, total and phosphorylated AKT, total and phosphorylated mTOR, and phospho-ERK1/2) immunohistochemistry
Time Frame: At study entry
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mutation Analysis
Description: To determine if relevant biomarkers correlate with response to treatment in each of the two arms. Unstained sections of tumor tissue and DNA extracted from whole blood will be used for mutational analysis (including PTEN, PIK3CA, KRAS, and CTNNB1 (beta-catenin) performed using a sequencing panel assay.
Time Frame: At study entry
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 30 days after the last cycle.
Description: Collected on a 28 day cycle while treatment continues and then up to 30 days after the last cycle.
Arm/Group | Everolimus and Letrozole | Tamoxifen and Medroxyprogesterone Acetate
All-Cause Mortality (participants affected / at risk) | 13/37 | 20/36
Serious Adverse Events (participants affected / at risk) | 13/37 | 10/36
Other Adverse Events (participants affected / at risk) | 37/37 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus and Letrozole (N=37) | Tamoxifen and Medroxyprogesterone Acetate (N=36)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Kidney Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0
Creatinine Increased (Investigations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms Benign, Malignant and Unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin and Subcutaneous Tissue Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus and Letrozole (N=37) | Tamoxifen and Medroxyprogesterone Acetate (N=36)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 25 | 20
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Heart Failure (Cardiac disorders) | 1 | 0
Cardiac Disorders - Other (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 1
Hearing Impaired (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Eye Disorders - Other (Eye disorders) | 1 | 1
Blurred Vision (Eye disorders) | 2 | 1
Vitreous Hemorrhage (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Dry Mouth (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 13 | 12
Diarrhea (Gastrointestinal disorders) | 18 | 7
Cheilitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 5
Bloating (Gastrointestinal disorders) | 1 | 2
Stomach Pain (Gastrointestinal disorders) | 1 | 0
Salivary Duct Inflammation (Gastrointestinal disorders) | 1 | 0
Rectal Mucositis (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 7 | 9
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Mucositis Oral (Gastrointestinal disorders) | 24 | 4
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 0
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 19 | 12
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 3
Lip Pain (Gastrointestinal disorders) | 1 | 0
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2
General Disorders And Administration Site Conditio (General disorders) | 0 | 1
Pain (General disorders) | 10 | 6
Malaise (General disorders) | 1 | 1
Localized Edema (General disorders) | 3 | 1
Flu Like Symptoms (General disorders) | 3 | 0
Non-Cardiac Chest Pain (General disorders) | 4 | 1
Edema Limbs (General disorders) | 15 | 9
Edema Face (General disorders) | 2 | 0
Fatigue (General disorders) | 22 | 15
Fever (General disorders) | 4 | 2
Chills (General disorders) | 4 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Infections And Infestations - Other (Infections and infestations) | 1 | 1
Wound Infection (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 0
Tooth Infection (Infections and infestations) | 2 | 0
Vulval Infection (Infections and infestations) | 2 | 0
Skin Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 1 | 1
Papulopustular Rash (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 1 | 0
Mucosal Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 5 | 1
Kidney Infection (Infections and infestations) | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0
Vaginal Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 6 | 1
Bronchial Infection (Infections and infestations) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Burn (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 1
Investigations - Other (Investigations) | 4 | 1
Weight Loss (Investigations) | 7 | 5
Weight Gain (Investigations) | 0 | 2
Platelet Count Decreased (Investigations) | 15 | 4
Lymphocyte Count Decreased (Investigations) | 4 | 2
Lipase Increased (Investigations) | 1 | 1
Inr Increased (Investigations) | 1 | 1
Creatinine Increased (Investigations) | 6 | 8
Cholesterol High (Investigations) | 16 | 3
Neutrophil Count Decreased (Investigations) | 12 | 3
Cd4 Lymphocytes Decreased (Investigations) | 2 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
White Blood Cell Decreased (Investigations) | 17 | 4
Aspartate Aminotransferase Increased (Investigations) | 14 | 8
Alkaline Phosphatase Increased (Investigations) | 7 | 1
Alanine Aminotransferase Increased (Investigations) | 11 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 7
Hyponatremia (Metabolism and nutrition disorders) | 4 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 8 | 1
Hypokalemia (Metabolism and nutrition disorders) | 13 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 | 12
Hypertriglyceridemia (Metabolism and nutrition disorders) | 20 | 8
Hypernatremia (Metabolism and nutrition disorders) | 5 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 23 | 11
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 13 | 8
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 5
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous System Disorders - Other (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 2
Stroke (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 5
Paresthesia (Nervous system disorders) | 2 | 1
Memory Impairment (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 15 | 3
Dysgeusia (Nervous system disorders) | 8 | 1
Syncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 3
Psychiatric Disorders - Other (Psychiatric disorders) | 1 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 9 | 4
Hallucinations (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 8 | 4
Delirium (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 5 | 4
Agitation (Psychiatric disorders) | 0 | 2
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 0 | 2
Urinary Urgency (Renal and urinary disorders) | 2 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 4 | 1
Urinary Tract Pain (Renal and urinary disorders) | 5 | 3
Urinary Frequency (Renal and urinary disorders) | 6 | 2
Renal Calculi (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 7 | 5
Hematuria (Renal and urinary disorders) | 2 | 2
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 0 | 1
Vaginal Pain (Reproductive system and breast disorders) | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 6
Perineal Pain (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 3
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 3
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 7
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 8 | 3
Nail Ridging (Skin and subcutaneous tissue disorders) | 3 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 3
Thromboembolic Event (Vascular disorders) | 1 | 5
Lymphedema (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 13 | 8
Hot Flashes (Vascular disorders) | 9 | 8
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02228681/Prot_SAP_000.pdf